CLINICAL TRIAL: NCT06834451
Title: Bioequivalence Study of Revolade® Eltrombopag 50 mg Tablets - Novartis Vs Myelone ® Eltrombopag 50 mg Tablets - Colompack / Immediate Release Tablets in Healthy Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Revolade® Eltrombopag 50 mg
Acronym: Eltrombopag
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Atencion e Investigacion Medica (Network)
Responsible Party: Principal Investigator, Humberto Reynales MD MSc PhD, Principla Investigator, Centro de Atencion e Investigacion Medica
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: ELTROM-BIO-001-2023
Record Dates: First submitted 2025-01-23; First posted 2025-02-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Healthy; Healthy Donors
Keywords: Bioequivalence
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Intervention Model Description: Bioequivalence study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Period 1 (Active Comparator): Revolade® Reference
  Interventions: Drug: Revolade®; Drug: Eltrombopag (EPAG)
- Period 2 (Active Comparator): Eltrombopag TEST
  Interventions: Drug: Revolade®; Drug: Eltrombopag (EPAG)

INTERVENTIONS:
Drug: Revolade® — Tableta 50 mg Reference
  Other Names: Eltrombopag
Drug: Eltrombopag (EPAG) — Tableta 50 mg

SUMMARY:
Bioequivalence Study

DETAILED DESCRIPTION:
A bioequivalence study of Eltrombopag will be developed in 30 healthy subjects, under fasting condition, following the design:

Open-label, crossover, randomized, single-dose design of 50 mg Eltrombopag tablets/immediate release tablets, with two treatments, two periods, two sequences in healthy volunteers in fasting condition, with a washout time of 15 days between each dose

ELIGIBILITY:
Inclusion Criteria:

* Women and men between 18 and 50 years of age. Have been clinically diagnosed as healthy by the trial physician. Subjects with clinical laboratory results requested in the protocol (Table 2) within normal ranges and/or fit by medical screening. Current for 3 months.

Subjects non-smokers for the last 3 months. Having signed the informed consent. Subjects sexually active or of reproductive age must use an effective contraceptive method during and for at least 7 days after the end of the study.

Body mass index between 18-30 kg/m2 at the time of inclusion in the study. Subject with complete contact information (cell phone and/or landline contact, address, email).

Subject who has a family member or guardian with a contact telephone number. Subject with the availability of time to comply with the scheduled visits and activities.

Exclusion Criteria:

* Subject with a diagnosis of renal, cardiac, hepatic, immunological, dermatological, endocrine, gastrointestinal, neurological or psychiatric disease.

Woman in a state of pregnancy or breastfeeding. Subject diagnosed with hematological disorders, such as anemias and/or polycythemia.

Subjects with a history of gastric surgeries. Permanent or temporary use during the last 15 days of any type of medication either on their own initiative or by medical prescription. Except female patients who are planning regularly with the same contraceptive method in the last 6 months prior to the start of the present trial.

Consumption of xanthines from coffee, tea or chocolate during the 48 hours prior to hospitalization.

Drinking alcohol in excess of 16 grams every week equivalent to 1 beer or 2 glasses of wine during the last 15 days prior to hospitalization.

Consumption of drugs of abuse or psychoactive substances reported as positive test at the time of hospitalization.

Known hypersensitivity to the active ingredient or excipients of the test product.

Medical history of angioedema or anaphylaxis. Subject diagnosed with human immunodeficiency virus infection, hepatitis B or hepatitis C positive.

Having participated in clinical studies in the 4 months prior to the time of signing the informed consent.

Having donated blood in the 30 days prior to the time of signing the informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Outcome Measures | 0- 6 hours
  Peak Plasma Concentration (Cmax)
Pharmacokinetic Outcome Measures | 0 - 6 hours
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atención e Investigación Médica, Chía, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Oct 2024 - Oct 2025
Access Criteria: Indicate whether a proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed
URL: https://www.caimed.com/